CLINICAL TRIAL: NCT07048626
Title: Impact of Low-Level Laser Therapy on Hair Regrowth Post PRP Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSAHSW/Batch-Fall23/903
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP treatment (Experimental)
  Interventions: Combination Product: PRP treatment
- low leve laser therapy post prp treatment (Active Comparator)
  Interventions: Combination Product: low level laser therapy post prp treatment

INTERVENTIONS:
Combination Product: PRP treatment — PRP treatment involves drawing a blood sample, processing it to concentrate platelets, and then injecting that concentrated plasma back into the body, typically at the site of an injury or area needing regeneration. The procedure aims to utilize the growth factors within the platelets to accelerate healing and tissue repair.
  Arms: PRP treatment
Combination Product: low level laser therapy post prp treatment — will receive low-level laser therapy post prp treatment upto 12 weeks .Low-level laser therapy (LLLT) is a non-invasive treatment for hair loss that uses low-intensity laser light to stimulate hair follicles and improve blood circulation. It's often used on its own or combined with other therapies like PRP.
  Arms: low leve laser therapy post prp treatment

SUMMARY:
Low-level laser stimulates cells in the hair follicles, which promotes hair growth. The patient's own blood platelets are used in platelet-rich plasma treatment to encourage hair growth. Combining low-level laser treatment with platelet-rich plasma will promote hair growth in patients.

DETAILED DESCRIPTION:
To determine the impact of low-level laser therapy on hair regrowth following prp treatment.

This will be case control study conducted on 22 participants with androgenetic alopecia (AGA).

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18-35 years diagnosed with androgenic alopecia or other non-scarring hair loss conditions.
* Having the Norwood-Hamilton scale placed in stages I-V for men Ludwig scale in stages I-III for women .

Exclusion Criteria:

* Use of systemic medications (e.g., corticosteroids, immunosuppressants) or treatments affecting hair regrowth within the last 3 months.
* History of hypersensitivity or adverse reactions to laser therapy
* Active systemic diseases such as uncontrolled diabetes, autoimmune disorders, or malignancies
* Pregnant or breastfeeding individuals.
* Patients with pacemakers or implanted medical devices contraindicated with low level laser therapy.
* History of hair transplant surgery in the treatment area

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Physician's Global Assessment (PGA) scale | 12 Months
  The Physician's Global Assessment (PGA) scale is a tool used by physicians to evaluate the overall severity of a patient's disease. It's a subjective assessment, typically on a scale of 0 to 3 or 0 to 4, with higher scores indicating more severe disease activity. The PGA focuses on the overall disease activity, considering both the severity of active manifestations and relevant laboratory results, excluding organ damage and subjective findings unrelated to disease activity

CONTACTS AND LOCATIONS:
Locations (1):
- Reshape Clinic, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No